CLINICAL TRIAL: NCT05990621
Title: A Single-arm, Open-label, Dose-escalation/Expansion, Early-phase Clinical Study of Anti-CD70 CAR-T Cell Injection in Patients With CD70-positive Advanced Urological Neoplasms
Brief Title: Anti-CD70 CAR-T Cell Injection in Patients With CD70-positive Advanced Urologic Neoplasms
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: UTC Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Anti-CD70 CAR-T Cell Injection
Record Dates: First submitted 2023-08-07; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: CD70-positive Advanced Urologic Neoplasms
Keywords: Anti-CD70 CAR-T; Urologic Neoplasms
MeSH Terms: conditions — Urologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Accelerated titration and 3+3 design dose escalation phase followed by dose expansion phase
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-CD70 CAR-T cells (Experimental): Anti-CD70 CAR-T cells are autologous genetically modified T cells.
  Interventions: Biological: Anti-CD70 CAR-T cells

INTERVENTIONS:
Biological: Anti-CD70 CAR-T cells — 0.6×106/Kg ～ 5.0×106/Kg; cells will be infused intravenously.

SUMMARY:
This is a single-arm, open-label, exploratory clinical study to evaluate the safety, tolerability and preliminary efficacy of Anti-CD70 CAR-T cell injection in patients with CD70-positive Advanced Urologic Neoplasms.

DETAILED DESCRIPTION:
This study will include two parts, dose escalation phase (accelerated titration and 3+3 design) followed by a dose expansion phase. All eligible participants will receive a conditioning chemotherapy regimen of fludarabine and cyclophosphamide followed by CAR-T cell injection.

The dose escalation phase will determine the maximum tolerated dose (MTD) of Anti-CD70 CAR-T cell injection. Additional patients will be enrolled in the dose expansion phase to further characterize the safety profile and evaluate the efficacy of Anti-CD70 CAR-T cell injection, and establish recommended phase 2 dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject is≥18 years old (including cut-off value), gender is not limited. 2. Histopathologically confirmed tumors of the urinary system (including renal cancers and urothelial cancers). Renal cancers should have failed after targeted therapy and/or immunotherapy. Urothelial cancers should have failed after chemotherapy and/or immunotherapy. Or subjects are unable to tolerate or lack effective therapies.

  3. At least one measurable lesion according to RECIST v1.1. 4. CD70 should be positive confirmed by Immunohistochemistry/Immunocytochemistry/ Flow Cytometry (IHC/ICC/FCM) in tumor tissue samples.

  5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. 6. Life expectancy ≥ 3 months. 7. Adequate function defined as: Hematological functions: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L (Patients should not receive G-CSF support within 7 days before laboratory examination); Absolute Lymphocyte Count (ALC) ≥ 0.5 × 109/L; Hemoglobin (HGB) ≥ 80 g/L (Patients should not be transfused red cells within 7 days before the laboratory examination); Platelet count (PLT) ≥ 75 × 109/L (Patients should not receive transfusion support within 7 days before the laboratory examination).

Hepatic functions: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 × upper limit of normal (ULN); AST and ALT of patients with liver metastasis ≤ 5 × ULN; Total bilirubin (TBIL) ≤ 1.5 × ULN; TBIL of patients with liver metastasis must ≤ 3.0 × ULN; TBIL of patients with Gilbert's Syndrome ≤ 3.0 × ULN and Direct bilirubin (DBIL) ≤ 1.5 × ULN.

Coagulation functions: International normalized ratio (INR) ≤ 1.5 × ULN; Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (Except for patients who are receiving therapeutic anticoagulants.).

Renal functions: Serum creatinine (Cr) ≤ 1.5 × ULN; or Estimated glomerular filtration rate (eGFR) ≥30ml/(min·1.73 m2)(Calculated by CKD⁃EPI).

Cardiac functions: Left ventricular ejection fraction (LVEF) > 50%; Pulmonary function: Oxygen saturation (SpO2) > 92%. 8. Female participants of childbearing potential must undergo a pregnancy test and the results must be negative. Female participants of childbearing potential or male participants whose sex partner has childbearing potential must be willing to use effective methods of contraception from screening period to at least 1 year after infusion.

9. Participants must be able to understand the protocol and be willing to enroll the study, sign the informed consent, and be able to comply with the study and follow-up procedures.

Exclusion Criteria:

* 1. Patients have received systemic therapy with cytotoxic chemicals, monoclonal antibodies, or immunotherapy within 4 weeks or 5 half-lives (which is shorter) prior to signing informed consent; Patients have received systemic glucocorticoids (prednisone at a dose of ≥10 mg per day or equivalent) or other immune-suppressive therapy within 2 weeks prior to signing informed consent; Patients have received systemic antitumor therapy with a biologic agent or other approved targeted small-molecule inhibitor within 1 week or five half-lives (which is shorter) prior to signing informed consent; Patients have received Chinese herbal medicine or Chinese patent medicine with anti-tumor indication within 1 week prior to signing informed consent.

  2. Pregnant or lactating women. 3. Patients with hepatitis B surface antigen (HBsAg) positive. Patients who is hepatitis B core antibody (HBcAb) positive and the quantification of HBV DNA in peripheral blood is higher than the lower limit of detection. Patients who is hepatitis C virus (HCV) antibody positive and quantification of HCV DNA in peripheral blood is higher than the lower limit of detection. Patients with human immunodeficiency virus (HIV) antibody positive. Patients with syphilis antibody positive and tolulized red unheated serum test (TRUST) titer ≥ 1:4.

  4. The toxicities caused by the prior therapy (surgery, chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc.) have not recovered to grade 1 according to CTCAE, except for hair loss and peripheral sensory nerve disorders.

  5. Have received any allogeneic tissue/organ transplantation (including bone marrow transplantation, stem cell transplantation, liver transplantation, kidney transplantation), except for the transplantation that does not require immunosuppressive therapy (such as: corneal transplantation, hair transplantation.) 6. Patients have received anti-CD70 CAR-T cell therapy. 7. Patients who have history of major surgery and unrecovered severe trauma within 4 weeks prior to signing informed consent; or plan to have major surgery within 12 weeks of cell therapy.

  8. Presence of known central nervous system metastases, but the following patients will be allowed: a) Asymptomatic brain metastases; b) Clinically stable (no radiographic progression within 4 weeks before apheresis and return of any neurologic symptoms to baseline), and with no need for corticosteroids or other treatment for brain metastases for ≥ 4 weeks.

  9. Patients with clinically significant systemic disease (such as: severe active infection or significant cardiac, pulmonary, hepatic, nervous system, or other organ dysfunction) that evaluated by the investigator would impair the patients' ability to tolerate the treatments used in this study or significantly increase the risk of complications.
  * Uncontrolled severe active infection (sepsis, bacteremia, viremia, etc.);
  * Congestive heart failure with New York Heart Association (NYHA) functional class > 1;
  * Clinically significant severe aortic stenosis and symptomatic mitral stenosis;
  * Electrocardiogram QTc > 450 msec or QTc > 480 msec in patients with bundle-branch block;
  * Uncontrolled clinically significant arrhythmia within 6 months prior to signing informed consent;
  * Acute coronary syndrome (such as: unstable angina, myocardial infarction) within 6 months prior to signing informed consent;
  * Drug-uncontrolled hypertension (systolic pressure ≥ 160 mmHg and/or diastolic pressure ≥ 100 mmHg) or pulmonary hypertension;
  * Cerebrovascular accident occurred within 6 months prior to signing informed consent, including transient ischemic attack (TIA), cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage;
  * A history of active, chronic, or recurrent (within 1 year prior to signing informed consent) severe autoimmune disease or immune-mediated disease requiring steroids or other immunosuppressive therapy, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel disease, Hashimoto's thyroiditis, autoimmune thyroid disease, multiple sclerosis. Exceptions: hypothyroidism that can be controlled only by hormone replacement therapy, skin diseases (such as: vitiligo, psoriasis) that do not require systemic treatment, coeliac disease that has been controlled; 10. Any form of primary or secondary immunodeficiency, such as severe combined immunodeficiency (SCID); 11. History of severe systemic hypersensitivity reaction to the drugs/ingredients [fludarabine, cyclophosphamide, dimethyl sulfoxide (DMSO), low molecular dextran, human serum albumin (HSA), etc.] used in this study.

    12. Patients have received attenuated vaccine within 4 weeks prior to signing informed consent.

    13. Patients have received other clinical trials within 4 weeks prior to signing informed consent.

    14. History of another malignancy tumor within the previous five years, except for adequately treated non-melanoma skin cancer, carcinoma in situ of bladder, stomach, colon, cervix/dysplasia, melanoma, or breast.

    15. History of neuropsychiatric diseases diagnosed by the ICD-11 criteria or evaluated by investigator, including but not limited to epilepsy, schizophrenia, dementia, drug and alcohol addictions.

    16. For any other reasons, the patients are believed not suitable for participation in this study by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | 2 years
  Incidence and severity of adverse events.
Serious Adverse Events (SAEs) | 2 years
  Incidence and severity of serious adverse events.
Adverse Events of Special Interest (AESI) | 2 years
  Incidence and severity of adverse event of special interest.
Identification of Maximum Tolerated Dose (MTD) | 4 weeks after the CAR-T cells infusion
  Incidence and severity of dose-limiting toxicities (DLTs) following infusion of UCL70802 cell injection, at each dose level tested in dose escalation phase.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  The Objective Response Rate (ORR) is the percentage of participants who achieved Complete Response (CR) or Partial Response (PR) based on RECIST version 1.1.
Duration of Overall Response (DOR) | 2 years
  Time from documentation of disease response to disease progression.
Progression-Free Survival (PFS) | 2 years
  PFS is defined as the time from CAR-T infusion to the date of the disease progression or death from any cause.
Overall Survival (OS) | 2 years
  OS is defined as the time from CAR-T infusion to the date of death due to any cause.
Bio-distribution of Anti-CD70 CAR-T cells | 2 years
  CAR copies will be measured by qPCR to evaluate the expansion and persistence of CAR-T cells in vivo.
Cytokine Level in Peripheral Blood | 2 years
  Level of cytokines (IFN-γ, IL-6, IL-2, etc.) in serum.
Number of participants with anti-drug antibodies. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Linhui Wang, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China